CLINICAL TRIAL: NCT06580561
Title: Move and Snooze: Adding Insomnia Treatment to an Exercise Program to Improve Pain Outcomes in Older Adults With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Whibley, Assistant Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00241352; 1R01AG081299-01A1 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis; Insomnia
Keywords: Exercise coaching; Cognitive behavioral therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized in blocks, stratified by biological sex, age, and baseline pain intensity (per protocol)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move and Snooze program (Experimental): This includes the personalized exercise program plus Cognitive Behavioral Therapy for Insomnia (CBT-I).
  Interventions: Behavioral: Personalized exercise coaching; Behavioral: Cognitive behavioral therapy for Insomnia
- Personalized exercise program (Experimental)
  Interventions: Behavioral: Personalized exercise coaching

INTERVENTIONS:
Behavioral: Personalized exercise coaching — This is a 6-session personalized exercise coaching program (delivered over 8 weeks).
  All participants will complete six 30-minute scheduled online or phone sessions with a health coach as part of a manualized personalized exercise program (once per week for the first four sessions and then once every two weeks for the remaining two sessions).
Behavioral: Cognitive behavioral therapy for Insomnia — This is a 6-week course of automated, digitally delivered cognitive behavioral therapy for insomnia delivered by the online program Sleepio. The weekly sessions will last approximately 15-20 minutes.
  Session content comprises evidence-based cognitive and behavioral techniques including Stimulus Control Therapy and Sleep Restriction Therapy, sleep hygiene education, and relaxation exercises.
  Arms: Move and Snooze program

SUMMARY:
This research will compare the effectiveness of a remotely delivered personalized exercise coaching plus an evidence-based sleep improvement intervention to remotely delivered personalized exercise coaching alone for knee osteoarthritis pain.

The study team hypothesize that the combined intervention will result in greater improvements in patient-reported pain intensity, recorded with real-time data capture, than remotely delivered exercise coaching alone.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported physician diagnosis of knee osteoarthritis
* Persistent knee osteoarthritis-related pain of at least moderate intensity (as indicated in the protocol)
* Indication of persistent symptoms of insomnia, determined by scoring on the Sleep Condition Indicator questionnaire (as indicated in the protocol)
* If receiving medication for pain or sleep disturbances, having had no change in prescription in the previous three months and be willing to make no other changes to medications for pain or sleep during the active study period.
* Adequate literacy level to ensure web-based surveys can be completed independently, as assessed using a brief 3-item literacy level screener

Exclusion Criteria:

* Concurrent diagnosis of a systemic, inflammatory musculoskeletal disorder (e.g., rheumatoid arthritis)
* Active malignancy
* Neurological conditions (e.g., movement disorders)
* Any medical condition which would make graded increase of physical activity unsuitable (determined by a positive answer to the question: "Has a doctor or healthcare professional advised you to avoid physical activity for any reason?").
* Unable to understand English sufficiently to take part in the intervention.
* Unable to provide electronic informed consent.
* Evidence of significant cognitive impairment (i.e., ≥2 errors on a 6-item cognitive screener).
* Presence of severe psychiatric disorder.
* Currently participating in an interventional trial or a pain or sleep management program or having done so in the past six months.
* Visual or hearing impairment that would prevent use of the intervention.
* Serious physical health concerns necessitating surgery or with a prognosis <6 months
* Irregular sleep-wake schedule, e.g., shift work.
* Self-report of diagnosis of a specific sleep disorder other than insomnia that is not currently adequately treated, e.g., sleep apnea or narcolepsy.
* Currently meeting or exceeding physical activity guidance from the U.S. Department of Health and Human Services (noted in protocol)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in average pain intensity using a 0-10 numerical rating scale between baseline and the 8-week follow-up (post-intervention) period | Baseline, 8-week follow-up (post-intervention)
  This is a one question numerical rating scale in which participants select from 0 (no pain) -10 (worst pain imaginable) numerical rating scale 4 times a day over 7 days during each assessment period (baseline and 8-week follow-up). These four within-day ratings collected over seven days will be averaged for each participant to provide a single pain intensity rating for each assessment period.

SECONDARY OUTCOMES:
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity 3a questionnaire between baseline and 8-week follow-up (post-intervention) | Baseline, 8-week (post-intervention)
  There are 3 questions that participants answer and from no pain (1) - very severe (5). There is a total score of 15 with a higher score indicating higher pain intensity.
Change in the PROMIS Pain Interference 8a questionnaire between baseline and 8-week follow-up (post-intervention) | Baseline, 8-week (post-intervention)
  There are 8 questions regarding the extent to which pain has interfered with activities over the past 7 days, ranging from not at all (1) - Very much (5). Total scores range from 8 to 40, with a higher score representing higher interference due to pain.
Change in the PROMIS Physical Function questionnaire between baseline and 8-week follow-up (post-intervention) | Baseline, 8-week (post-intervention)
  There are 4 questions regarding function that participants answer and from without any difficulty (5) - unable to do (1). And 4 questions for that participants select from not at all (5) to cannot do (1). There is a total score of 40 with a higher score indicating greater physical function.
Change in the Quality of Life subscale of the Knee injury and Osteoarthritis Outcome Score (KOOS) between baseline and 8-week follow-up (post-intervention) | Baseline, 8-week (post-intervention)
  The KOOS quality of life subscale includes 4 questions. The Score subscale is scored using a Likert scale with five possible answers, ranging from 0 (no problems) to 4 (extreme problems). The quality of life subscale score is then normalized to a 0-100 scale, with higher scores equaling better status. 0 represents extreme knee problems and 100 represents no knee problems.
Patient Global Impression of Change at 8-week follow-up (post-intervention) | 8-week (post-intervention)
  This is a one question survey that participants will select from very much improved (1) -very much worse (7) since the start of the study and overall status. A lower number indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Whibley, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data will be transmitted to and stored at the Inter-university Consortium for Political and Social Research data repository.
Supporting Information: Study Protocol, ICF
Time Frame: Final submission and release of the study data will occur approximately 8 and 12 months following the end of fieldwork, respectively, and within the award period. Study data deposited in the Inter-university Consortium for Political and Social Research data repository will be available to the research community in perpetuity.
Access Criteria: Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the Inter-university Consortium for Political and Social Research data repository.
URL: https://www.icpsr.umich.edu/web/pages/